CLINICAL TRIAL: NCT06989515
Title: Does Anejaculation Reflect Better Clinical Outcomes in BPO Patients Receiving Silodosin?
Brief Title: Clinical Outcomes and Ejaculatory Function in BPO Patients Treated With Silodosin
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tarik Emre Sener, Assoc. Prof., Marmara University
Other Study IDs: MAR.UAD.0023
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostate Obstruction (BPO); Lower Urinary Tract Symptom; Ejaculatory Dysfunction; Anejaculation; Silodosin
Keywords: Silodosin; Ejaculatory Dysfunction; Benign Prostatic Obstruction; Lower Urinary Tract Symptoms; Alpha-blocker Side Effects
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Ejaculatory Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anejaculation: Male patients who develop anejaculation after initiating silodosin treatment for benign prostatic obstruction (BPO).
- Non-Anejaculation: Male patients who do not develop anejaculation during silodosin treatment for benign prostatic obstruction (BPO).

SUMMARY:
This observational study aims to evaluate the relationship between silodosin-induced anejaculation and clinical outcomes in male patients with benign prostatic obstruction (BPO). Silodosin is a commonly used alpha-blocker for lower urinary tract symptoms (LUTS). However, it may cause ejaculatory dysfunction, particularly anejaculation. In this study, patients receiving silodosin for the first time will be grouped based on whether they experience anejaculation or not. Treatment response will be assessed using urinary flow rate, post-void residual urine, and International Prostate Symptom Score (IPSS). Sexual function will be evaluated using the International Index of Erectile Function-5 (IIEF-5) before and after treatment. The study aims to explore whether the presence of anejaculation is associated with improved symptom relief or differences in sexual health.

DETAILED DESCRIPTION:
This is a observational study designed to investigate the association between silodosin-induced anejaculation and clinical outcomes in patients diagnosed with benign prostatic obstruction (BPO). Silodosin is an alpha-1A adrenergic receptor antagonist frequently used in the treatment of lower urinary tract symptoms (LUTS) secondary to BPO. One of the common adverse effects of silodosin is ejaculatory dysfunction, particularly anejaculation or retrograde ejaculation.

In this study, male patients over 40 years of age who are newly prescribed silodosin (8 mg/day) for LUTS will be enrolled. Baseline assessments will include serum PSA levels, prostate volume measurement via ultrasonography, uroflowmetry, post-void residual (PVR) urine volume, the International Prostate Symptom Score (IPSS), and the International Index of Erectile Function-5 (IIEF-5). These assessments will be repeated at the first routine follow-up visit, approximately one month after treatment initiation.

Patients will be divided into two groups based on the presence or absence of anejaculation. The primary objective is to compare changes in LUTS-related parameters (IPSS, uroflowmetry, PVR) and erectile function (IIEF-5 scores) between the two groups. This study will help determine whether anejaculation, a common side effect of silodosin, correlates with improved therapeutic response or changes in sexual health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 40 years or older
* Diagnosed with lower urinary tract symptoms (LUTS) due to benign prostatic obstruction (BPO)
* Initiating silodosin 8 mg/day therapy for the first time
* Able to complete IPSS and IIEF-5 questionnaires
* Willing and able to provide written informed consent

Exclusion Criteria:

* History of prior treatment with silodosin or other α-blockers in the last 3 months
* Known neurogenic bladder or history of neurological disease affecting voiding
* History of prostate surgery or pelvic radiation
* Diagnosed prostate or bladder malignancy
* Use of medications affecting sexual function (e.g., PDE5 inhibitors) within the last month
* Severe cardiovascular, hepatic, or renal comorbidities
* Cognitive impairment preventing informed consent or questionnaire completion

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients aged 40 years and older presenting with lower urinary tract symptoms due to benign prostatic obstruction (BPO), who are newly prescribed silodosin therapy and have no prior history of prostate surgery or neurogenic bladder dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) | Baseline and 1 Month
  IPSS will be measured at baseline and after 1 month of silodosin therapy. The change in score will be compared between patients who develop anejaculation and those who do not.
Change in Maximum Urinary Flow Rate (Qmax) | Baseline and 1 Month
  Qmax will be measured via uroflowmetry at baseline and 1 month. Changes will be compared between the two groups.

SECONDARY OUTCOMES:
Change in Erectile Function (IIEF-5 Score) | Baseline and 1 Month
  Erectile function will be assessed using the IIEF-5 questionnaire at baseline and at 1 month. Changes will be compared between groups.
Change in Post-Void Residual Urine Volume (PVR) | Baseline and 1 Month
  PVR volume will be measured by ultrasonography at baseline and at 1 month. Changes will be analyzed between patients with and without anejaculation.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to privacy concerns and institutional data protection policies. However, access to anonymized data may be considered upon reasonable scientific request, subject to ethical approval and data sharing agreements.